CLINICAL TRIAL: NCT02574728
Title: AflacST1502: A Phase II Study of Sirolimus in Combination With Metronomic Chemotherapy in Children With Recurrent and/or Refractory Solid and CNS Tumors
Brief Title: Sirolimus in Combination With Metronomic Chemotherapy in Children With Recurrent and/or Refractory Solid and CNS Tumors
Acronym: AflacST1502
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Cannonball Kids' Cancer Foundation (Other); Hyundai Hope On Wheels (Other)
Responsible Party: Principal Investigator, William T Cash, Associate Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00082488
Record Dates: First submitted 2015-10-02; First posted 2015-10-14 (Estimated); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Cancer
Keywords: Pediatrics; Brain Tumors; Medulloblastoma; Ependymoma; Atypical teratoid rhabdoid tumor (ATRT); Pineoblastoma; Germ cell tumors (CNS and non-CNS); Neuroblastoma; Osteosarcoma; Ewing's Sarcoma; Rhabdomyosarcoma; Wilms Tumors; Soft Tissue Sarcomas; Langerhans cell histiocytosis (LCH); Histiocytic disorders; Rare pediatric solid tumors; Carcinomas
MeSH Terms: conditions — Neoplasms; Brain Neoplasms; Medulloblastoma; Ependymoma; Rhabdoid Tumor; Pinealoma; Neoplasms, Germ Cell and Embryonal; Neuroblastoma; Osteosarcoma; Sarcoma, Ewing; Rhabdomyosarcoma; Sarcoma; Histiocytosis, Langerhans-Cell; Carcinoma | interventions — Sirolimus; Celecoxib; Etoposide; etoposide phosphate; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Oral sirolimus, celecoxib, etoposide, and cyclophosphamide (Experimental): Participants in this group will receive oral sirolimus and celecoxib in addition to cycles of oral etoposide and cyclophosphamide for up to two years.
  Interventions: Drug: Sirolimus; Drug: Celecoxib; Drug: Etoposide; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Sirolimus — The starting dose for sirolimus is 2 mg/m2 once daily. The dose of sirolimus will be individually adjusted to achieve a target serum trough concentration in the range of 10-15 ng/ml. Sirolimus will be given by mouth every day for six weeks (every six weeks is called one cycle) for up to two years or 16 cycles.
  Other Names: Rapamune; rapamycin
Drug: Celecoxib — Celecoxib 100 mg will be given by mouth twice a day for six weeks (every six weeks is called one cycle) for up to two years or 16 cycles.
Drug: Etoposide — Etoposide 50 mg/m2 (maximum dose 100 mg) will be given daily by mouth for the first 3 weeks of a 6 week cycle. Six week cycles will be repeated for up to two years or 16 cycles.
  Other Names: Etopophos; Toposar
Drug: Cyclophosphamide — Cyclophosphamide 2.5 mg/Kg (maximum dose 100 mg) will be given daily by mouth for the second 3 weeks of a 6 week cycle. Six week cycles will be repeated for up to two years or 16 cycles.
  Other Names: Cytoxan

SUMMARY:
This study aims to determine the efficacy of daily sirolimus and celecoxib, with low dose etoposide alternating with cyclophosphamide for pediatric participants with relapsed or refractory tumors.

DETAILED DESCRIPTION:
This study aims to learn if the combination of oral sirolimus once daily with celecoxib, and with oral etoposide alternating every 21 days with oral cyclophosphamide (metronomic chemotherapy) is effective in shrinking relapsed or refractory tumors in pediatric participants. In addition, this study seeks to learn the length of time this combination can keep the tumor from growing, learn more about the side effects of sirolimus when used in this combination, and to learn if the sirolimus is working by evaluating blood and tumor tissue.

ELIGIBILITY:
Inclusion Criteria:

* Participants with any of the following tumors who have experienced relapse following front-line therapy, or who are refractory to front-line therapy, and participants with tumors that carry a poor prognosis and have no known standard curative therapy

  * Brain tumors of all World Health Organization (WHO) grades, except diffuse intrinsic pontine glioma (DIPG) - enrollment in the brain tumor stratum is closed
  * Extracranial solid tumors including histiocytoses
* Participants must have had a histologic verification of malignancy at original diagnosis or relapse, except in participants with optic pathway gliomas, or participants with pineal tumors and elevations of serum or cerebrospinal fluid (CSF) alpha-fetoprotein (AFP) or beta-human chorionic gonadotropin (beta-HCG)
* Tissue blocks or slides must be sent
* Participants must have radiographically measurable disease at the time of study enrollment to be eligible. Patients with neuroblastoma who do not have measurable disease but have metaiodobenzylguanidine (MIBG+) evaluable disease are eligible. Measurable disease in patients with CNS involvement is defined as tumor that is measurable (≥ 10 mm) in two perpendicular diameters on MRI and visible on more than one slice. For all patients, tumors that are located in a previously irradiated area may be considered measurable if the lesion has shown tumor growth after radiation or has been biopsied and proven to have active disease.
* Participant's current disease state must be one for which there is no known curative therapy
* Karnofsky performance level of greater than or equal to 50 percent for participants who are greater than 16 years of age at the time of screening
* Lansky performance level of greater than or equal to 50 percent for participants who are less than or equal to 16 years of age at the time of screening
* Fully recovered from acute toxic effects of all prior anti-cancer therapy
* Adequate bone marrow function as deemed by the protocol at the time of screening
* Adequate renal function as deemed by the study protocol at the time of screening
* Adequate liver function as deemed by the study protocol at the time of screening
* Serum triglyceride level ≤300 mg/dL and serum cholesterol ≤ 300 mg/dL
* Random or fasting blood glucose within the upper normal limits for age
* Adequate pulmonary function as deemed by the study protocol at the time of screening

Exclusion Criteria:

* Women who are currently pregnant or breastfeeding
* Receiving corticosteroids who have not been on a stable dose for at least 7 days
* Currently receiving enzyme inducing anticonvulsants
* Currently receiving receiving potent CYP3A4 (enzyme) inducers or inhibitors
* Currently receiving another investigational drug
* Currently receiving any other anti-cancer agents
* The use of cannabis oil is prohibited during the first 2 cycles of this protocol. Patients must be off of cannabis oil for 3 days prior to enrollment.
* Uncontrolled infection
* Participants who in the opinion of the investigator may not be able to comply with the safety monitoring requirements

Ages: 12 Months to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 46 (Actual)
Dates: Start 2015-06; Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Radiographic response to treatment for solid tumors | Baseline, End of Treatment (Up to 2 years)
  Radiographic response to treatment will be assessed by Response Evaluation Criteria in Solid Tumors (RECIST) for participants with solid tumors via CT or MRI scan. A complete response (CR) is a disappearance of all target and non-target lesions. Partial response (PR) is at least a 30% decrease in the disease measurement compared to the baseline measurement. Stable disease (SD) is neither sufficient shrinkage to qualify for partial response (PR) nor sufficient increase to qualify for progressive disease (PD) taking as reference the smallest disease measurement since baseline. Progressive disease (PD) is at least a 20% increase in the disease measurement compared to baseline, or the appearance of one or more new lesions, or evidence of laboratory or clinical progression.
Radiographic response to treatment for central nervous system (CNS) tumors | Baseline, End of Treatment (Up to 2 years)
  Radiographic response to treatment will be assessed for participants with CNS tumors via CT or MRI scan. Response criteria are assessed based on the lesion of the longest diameter and its longest perpendicular diameter. Development of new disease or progression in any established lesions is considered progressive disease, regardless of response in other lesions. Complete response (CR) is the the disappearance of all target lesions. Partial response (PR) is greater than or equal to 50% decrease decrease in the sum of the products of the two perpendicular diameters of all target lesions, taking into reference the baseline measurement. Stable disease (SD) is neither a sufficient decrease in the sum of the products of the two perpendicular diameters of all target lesions to qualify for PR, nor sufficient increase in a single target lesion to qualify for progressive disease (PD).

SECONDARY OUTCOMES:
Number of adverse events | Baseline, End of Treatment (Up to 2 years)
  The adverse events associated with sirolimus in combination with metronomic chemotherapy administered on this schedule will be defined and evaluated throughout the treatment period.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Cash, MD, Principal Investigator — Emory University
Locations (6):
- United States (6):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Nemours/Alfred I. duPont Hospital for Children, Wilmington, Delaware
  - Children's Healthcare of Atlanta-Egleston, Atlanta, Georgia
  - Children's Healthcare of Atlanta, Scottish Rite, Atlanta, Georgia
  - Children's Mercy Hospital, Kansas City, Missouri
  - University of Virginia Health System, Charlottesville, Virginia